CLINICAL TRIAL: NCT06166732
Title: The Effect of Music-Based Mindfulness on Acculturative Stress and Attention in East Asian International Students
Brief Title: The Effect of Music-Based Mindfulness to Cope with Acculturative-Related Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Teresa Lesiuk, Professor, University of Miami
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20231114
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Stress
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Music-based Mindfulness Group (Experimental): Participants will receive a music-based mindfulness for 20 minutes.
  Interventions: Behavioral: Music-based Mindfulness
- Control Group (Other): Participants will receive a information session for 20 minutes.
  Interventions: Behavioral: Control Group

INTERVENTIONS:
Behavioral: Music-based Mindfulness — The participants will receive a single 20-minute music-based mindfulness session in person. The participants will listen to instrumental music during the session.
  Arms: Music-based Mindfulness Group
Behavioral: Control Group — The participants will receive a single 20-minute information session in person. The information session will introduce the definition, history, basic concepts, and benefits of mindfulness practice.
  Arms: Control Group

SUMMARY:
The purpose of this study is to explore the effect of music-based mindfulness on stress reduction among East Asian international students.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years of age or older
* Pursuing an undergraduate/graduate degree with an F-1 visa
* Originating from regions including China, Hong Kong, Taiwan, North Korea, South Korea, and Japan
* Living in the United States for no more than 3 years
* Having less than one year of mindfulness practice

Exclusion Criteria:

• Individuals not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2024-02-17 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Change in Spielberger State-Anxiety Inventory | 5 minutes before intervention and 5 minutes post intervention
  The Spielberger State-Trait Anxiety Inventory survey which has six-item short-form of the state(STAI: Y-6 score.
  To calculate the total STAI score (range 20 - 80):
  * reverse scoring of the positive items (calm, relaxed, content) so 1=4, 2=3, 3=2 and 4=1;
  * sum all six scores;
  * multiply total score by 20/6;
  * refer to Spielberger's manuals to interpret scores (a 'normal' score is approx. 34 - 36) Participant will complete the survey 5 minutes prior to the intervention and then 5 minutes after the intervention
Change in researcher-designed attention scale | 5 minutes before intervention and 5 minutes post intervention
  There are two items. The first item "I am very focused in the present right now" will utilize a 5-point scale ranging from 1= "Not at All" to 5= "Extremely." Conversely, the second item "I have a lot of distracting thoughts right now" will be measured using a reversed score. In this context, higher scores signify greater levels of attention. A composite score of these two items will be reported.
Change in Trail Making Test, Part A and B | 5 minutes before intervention and 5 minutes post intervention
  The Trail Making Test (TMT) is a timed test and the goal is to complete the test as accurately and as quickly as possible. Raw scores are reported in seconds to complete the test. For Part B, an average score is 75 seconds and a deficient score is greater than 273 seconds.
  The present study reports T-scores, which can range from a minimum of 0 and a maximum of 100. The higher the T- score achieved by a participant, the better the performance, indicating a higher level of functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Lesiuk, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Volpe 206, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No